CLINICAL TRIAL: NCT01404481
Title: Clean Intermittant Self Catheterisation: A Randomised Control Trial Comparing Single Use vs Reuse of Nelaton Catheters
Brief Title: Clean Intermittant Self Catheterisation: A Trial Comparing Single Use vs Reuse of Nelaton Catheters
Acronym: SURE
Status: Completed | Type: Observational
Sponsor: St George Hospital, Australia (Other)
Responsible Party: Principal Investigator, Hayley Leek, Hayley Leek CNS Urology/Continence NCA, St George Hospital, Australia
Other Study IDs: 09/STG/176
Record Dates: First submitted 2011-07-27; First posted 2011-07-28 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Urinary Retention
Keywords: Urinary retention; CISC; Single use; Re use
MeSH Terms: conditions — Urinary Retention | interventions — Catheters

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Single use group: New catheter for each Clean Intermittent Self Catheterisation (CISC), then discard.
  Interventions: Device: clean intermittent self catheterisation single use vs re use
- Re use of catheters group: Use same catheter for 1week- Cleaning with sunlight liquid soap, air dry or dry with lint free towel, store in a snap lock bag.
  Discard catheter and snap lock bag at end of each week.
  Interventions: Device: clean intermittent self catheterisation single use vs re use

INTERVENTIONS:
Device: clean intermittent self catheterisation single use vs re use — Over the 16 week period all patient will participate in 8 weeks of single use cathetersation and 8 weeks of re use catheterisation. The study is a randomised control crossover trial
  Other Names: Nelaton; Catheters

SUMMARY:
The purpose of the study is to compare single use of catheters with reuse of catheters for intermittant self catheterisation.

DETAILED DESCRIPTION:
Patients with voiding dysfunction and chronic urinary retention are taught the technique Clean Intermittent Self Catheterisation (CISC) by specialist Nurse Continence Advisors.

For several decades, patients have been taught to catheterise using a "clean" technique where they rinse their catheter under tap water and store the catheter in a sterile solution (e.g. Milton). The catheter is re-used for up to one week. The risk of urinary tract infection (UTI) was known to be minimal (and certainly much less than having a permanent indwelling catheter).

Recently, the Therapeutics Goods Administration has issued a guideline that CISC catheters should be "single-use items" but no data to support this guideline appears to have been collected.

The aim of this project is to assess the incidence of urinary tract infection (UTI) when comparing single-use catheters with re-use of catheters for CISC, and to determine the cost differences between the two methods.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* CISC > 2/day
* No current symptomatic UTI
* Willing to change catheter use method

Exclusion Criteria:

* Symptomatic Urinary Tract infection despite treatment
* <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Continence clinic, community patients, hospital patients
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2010-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Rate of Urinary Tract Infection | 16 weeks
  Urine specimens are sent at 4 weekly intervals over 16 weeks to check for Urinary tract infection

SECONDARY OUTCOMES:
Economic Cost | 16 weeks
  Difference in econimic cost of single use Catheterisation and re use catheterisation and the impact on the patient

CONTACTS AND LOCATIONS:
Overall Officials: Kate Moore, A/Professor, Principal Investigator — St George Hospital; Dr Emmanuel Karantanis, Doctor, Principal Investigator — St George Hospital
Locations (1):
- Pelvic Floor Bladder Unit St George Hospital, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Prieto JA, Murphy CL, Stewart F, Fader M. Intermittent catheter techniques, strategies and designs for managing long-term bladder conditions. Cochrane Database Syst Rev. 2021 Oct 26;10(10):CD006008. doi: 10.1002/14651858.CD006008.pub5. PMID 34699062